CLINICAL TRIAL: NCT00784238
Title: An Open-label, Prospective, Non-Comparative Study to Evaluate Subjective Well-Being and Responses in Patients With Schizophrenia Who Had Switched to Paliperidone Extended-Release Tablets
Brief Title: Efficacy Study of Paliperidone to Evaluate Subjective Change in Well-being and Drug Attitude in Schizophrenic Participants
Acronym: Power
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015391; R076477SCH4028
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Results first posted 2014-03-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone Extended-release; Paliperidone; R076477
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone (Experimental): Paliperidone Extended-Release (ER) oral tablet will be administered once daily at a starting dose of 6 milligram (mg) for 24 weeks, wherein dose range will be 3 to 12 mg per day.
  Interventions: Drug: Paliperidone

INTERVENTIONS:
Drug: Paliperidone — Paliperidone ER oral tablet will be administered once daily at a starting dose of 6 milligram (mg) for 24 weeks, wherein dose range will be 3 to 12 mg per day.
  Other Names: R076477; Invega Extended-release tablet

SUMMARY:
The purpose of this study is to evaluate improvement and efficacy of paliperidone extended-release for subjective well-being and drug attitudes of participants, when switching from oral antipsychotics in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-centric (conducted in more than one center), prospective (study following participants forward in time), and non-comparative study, in participants with schizophrenia. The study consists of following parts: Screening (that is, 14 days before study commences on Day 1); Acute Treatment phase (24 weeks); Extension phase 1 (24 weeks), which will be followed by additional Extension phase 2 (48 weeks). Total study duration per participant will be 96 weeks. Efficacy will primarily be evaluated by change from Baseline in Subjective Well-being Under Neuroleptic (SWN-20) Scale score and change from Baseline in Drug Attitude Inventory scores. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are diagnosed with schizophrenia (diagnosis criteria: Diagnostic and Statistical Manual of Mental Disorders, fourth edition [DSM-IV])
* Participants who need to change the antipsychotic drug to another one for the following reasons among the participants treated with an antipsychotic drug for more than two weeks before the screening-Lack of efficacy, lack of tolerance or lack of compliance
* Participants who are capable of and willing to fill out the questionnaire for themselves
* Childbearing potential women who consent to the use of the consistently permissible contraception (oral contraceptive, contraceptive injection, intrauterine device, double barrier method and contraceptive patch)
* Participants who are compliant with self-medication or can receive consistent help or support

Exclusion Criteria:

* Participants with the past history of neuroleptic malignant syndrome (NMS), or with allergy or hypersensitivity to risperidone or paliperidone
* Participants who have taken clozapine within one month before screening
* Participants who are suspicious of having clinically significant risk including suicide or aggressive behavior and are expected to unable to complete the study (based on the investigator's judgment)
* Participants with severe preexisting gastrointestinal narrowing (pathologic or iatrogenic) or participants who cannot swallow the drug whole (The study drug must not be chewed, divided, melted or grinded because it can impact the study drug release profile)
* Participants with a known or suspected history (for 6 months and longer) of substance dependence according to the DSM-IV criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (11):
- South Korea (11):
  - Busan
  - Changnyeong
  - Chungcheongbuk-Do
  - Daegu
  - Daejeon
  - Hwasun Gun
  - Iksan
  - Jeonju
  - Junam
  - Kwangjoo
  - Naju

REFERENCES:
- [Derived] Kim SW, Yoon JS, Kim YS, Ahn YM, Kim CE, Go HJ, Chee IS, Jung SW, Chung YC, Kim YD, Joe S, Lee J, Kwon YJ, Yoon BH, Jae YM. The effect of paliperidone extended release on subjective well-being and responses in patients with schizophrenia. Prog Neuropsychopharmacol Biol Psychiatry. 2012 Aug 7;38(2):228-35. doi: 10.1016/j.pnpbp.2012.04.004. Epub 2012 Apr 10. PMID 22516251

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone: Paliperidone Extended-Release (ER) oral tablet was administered once daily at a starting dose of 6 milligram (mg) for 24 weeks, wherein dose range was 3 to 12 mg per day.
Period: Overall Study
Arm/Group | Paliperidone
Started | 289
Completed | 170
Not Completed | 119
Not completed — Adverse Event | 14
Not completed — Death | 2
Not completed — Lack of Efficacy | 33
Not completed — Lost to Follow-up | 29
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 26
Not completed — Other | 14

BASELINE CHARACTERISTICS:
Arm/Group | Paliperidone
Number analyzed (Participants) | 289
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153
  Male | 136

OUTCOME MEASURES:

1. Primary Outcome: Subjective Well-being Under Neuroleptic (SWN-20) Scale Total Score at Week 24
Description: The SWN-20 scale is a 20 item scale that was originally designed to explore the subjective experience of psychotic participants. The SWN scale contains five sub-scales consisting of four items each: mental functioning (MF), self-control (SC), emotional regulation (ER), and social integration (SI), physical functioning (PF). The total score ranges from a minimum of 20 (poor subjective experience) to a maximum of 120 (excellent subjective experience). SWN scores appear to correlate with measure of objective psychopathology, quality of life and other self-ratings of mood.
Time Frame: Week 24
Population: Intent to treat (ITT) population for efficacy included all the participants who received paliperidone extended-release (ER) at least once and who had at least 1 post baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone
Number analyzed (Participants) | 284
Units on a scale | 77.89 (17.95)

2. Primary Outcome: Change From Baseline in Subjective Well-being Under Neuroleptic (SWN-20) Scale at Week 24
Description: The SWN-20 scale is a 20 item scale that was originally designed to explore the subjective experience of psychotic participants. The SWN scale contains five sub-scales consisting of four items each: mental functioning (MF), self-control (SC), emotional regulation (ER), and social integration (SI), physical functioning (PF). The total score ranges from a minimum of 20 (poor subjective experience) to a maximum of 120 (excellent subjective experience). SWN scores appear to correlate with measure of objective psychopathology, quality of life and other self-ratings of mood. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: The ITT population for efficacy included all the participants who received paliperidone ER at least once and who had at least 1 post baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Paliperidone (Lack of Efficacy Group): Paliperidone ER tablet at a dose ranging from 3 to 12 milligram (mg) per day was given orally for 24 weeks as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics for the main reason of lack of efficacy (switching of antipsychotic drug was clinically necessary because of no or insufficient response to treatment despite antipsychotic drug therapy at an adequate dose).
- Paliperidone (Lack of Tolerability Group): Paliperidone ER tablet at a dose ranging from 3 to 12 mg per day was given orally for 6 months as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics for the main reason of lack of tolerability (switching of antipsychotic drug was necessary due to lack of tolerability or safety problem in the existing antipsychotic drug).
- Paliperidone (Lack of Compliance Group): Paliperidone ER tablet at a dose ranging from 3 to 12 mg per day was given orally for 6 months as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics for the main reason of lack of compliance (switching of antipsychotic drug was necessary due to lack of compliance in the existing antipsychotic drug).
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 179 | 47 | 58
Units on a scale
  Baseline | 74.59 (17.81) | 76.51 (17.61) | 81.19 (15.68)
  Change at Week 24 | -1.59 (13.75) | -2.66 (13.72) | -0.93 (16.93)

3. Primary Outcome: Change From Baseline in Mental Functioning Subscale Score Based on Subjective Well-being Under Neuroleptic (SWN-20) Scale at Week 24
Description: The SWN-20 scale is a 20 item scale that was originally designed to explore the subjective experience of psychotic participants. The SWN scale contains five sub-scales consisting of four items each: mental functioning (MF), self-control (SC), emotional regulation (ER), and social integration (SI), physical functioning (PF). The total score ranges from a minimum of 20 (poor subjective experience) to a maximum of 120 (excellent subjective experience). SWN scores appear to correlate with measure of objective psychopathology, quality of life and other self-ratings of mood. Mental functioning subscale score ranges from 0 to 24 and higher score indicates improvement of disease. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 179 | 47 | 58
Units on a scale | -0.14 (3.56) | -0.51 (3.62) | -0.24 (4.79)

4. Primary Outcome: Change From Baseline in Self-Control Subscale Score Based on Subjective Well-being Under Neuroleptic (SWN-20) Scale at Week 24
Description: The SWN-20 scale is a 20 item scale that was originally designed to explore the subjective experience of psychotic participants. The SWN scale contains five sub-scales consisting of four items each: mental functioning (MF), self-control (SC), emotional regulation (ER), and social integration (SI), physical functioning (PF). The total score ranges from a minimum of 20 (poor subjective experience) to a maximum of 120 (excellent subjective experience). SWN scores appear to correlate with measure of objective psychopathology, quality of life and other self-ratings of mood. Self-Control subscale score ranges from 0 to 24 and higher score indicates improvement of disease. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 179 | 47 | 58
Units on a scale | -0.72 (3.74) | -0.62 (4.05) | -0.29 (4.07)

5. Primary Outcome: Change From Baseline in Emotional Regulation Subscale Score Based on Subjective Well-being Under Neuroleptic (SWN-20) Scale at Week 24
Description: The SWN-20 scale is a 20 item scale that was originally designed to explore the subjective experience of psychotic participants. The SWN scale contains five sub-scales consisting of four items each: mental functioning (MF), self-control (SC), emotional regulation (ER), and social integration (SI), physical functioning (PF). The total score ranges from a minimum of 20 (poor subjective experience) to a maximum of 120 (excellent subjective experience). SWN scores appear to correlate with measure of objective psychopathology, quality of life and other self-ratings of mood. Emotional Regulation subscale score ranges from 0 to 24 and higher score indicates improvement of disease. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 179 | 47 | 58
Units on a scale | -0.07 (3.61) | 0.11 (4.07) | 0.45 (3.97)

6. Primary Outcome: Change From Baseline in Physical Functioning Subscale Score Based on Subjective Well-being Under Neuroleptic (SWN-20) Scale at Week 24
Description: The SWN-20 scale is a 20 item scale that was originally designed to explore the subjective experience of psychotic participants. The SWN scale contains five sub-scales consisting of four items each: mental functioning (MF), self-control (SC), emotional regulation (ER), and social integration (SI), physical functioning (PF). The total score ranges from a minimum of 20 (poor subjective experience) to a maximum of 120 (excellent subjective experience). SWN scores appear to correlate with measure of objective psychopathology, quality of life and other self-ratings of mood. Physical Functioning subscale score ranges from 0 to 24 and higher score indicates improvement of disease. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 179 | 47 | 58
Units on a scale | -0.11 (4.15) | -0.68 (4.25) | 0.47 (4.50)

7. Primary Outcome: Change From Baseline in Social Integration Subscale Score Based on Subjective Well-being Under Neuroleptic (SWN-20) Scale at Week 24
Description: The SWN-20 scale is a 20 item scale that was originally designed to explore the subjective experience of psychotic participants. The SWN scale contains five sub-scales consisting of four items each: mental functioning (MF), self-control (SC), emotional regulation (ER), and social integration (SI), physical functioning (PF). The total score ranges from a minimum of 20 (poor subjective experience) to a maximum of 120 (excellent subjective experience). SWN scores appear to correlate with measure of objective psychopathology, quality of life and other self-ratings of mood. Social integration subscale score ranges from 0 to 24 and higher score indicates improvement of disease. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 179 | 47 | 58
Units on a scale | -0.55 (3.33) | -0.96 (3.26) | -1.31 (4.04)

8. Primary Outcome: Drug Attitude Inventory (DAI-10) Total Score at Week 24
Description: The DAI-10 is a 10-item questionnaire to assess 1) subjective experience of drug and 2) attitudes and beliefs toward neuroleptics which may influence compliance in schizophrenia participants. It is the binary scale assessing the participant's subjective response. A 'compliant' response is scored as +1; a dysphoric response is scored as -1. A positive sum of items indicates a positive subjective response (SR); a negative sum of scores indicates a negative SR (non-compliant). The final score is the grand total of the positive and negative points. Total score ranges from (-) 10 to (+) 10, higher score indicates positive SR (compliant) and lower score indicates negative SR (non-compliant).
Time Frame: Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone
Number analyzed (Participants) | 284
Units on a scale | 3.58 (4.73)

9. Primary Outcome: Change From Baseline in Drug Attitude Inventory (DAI-10) at Week 24
Description: The DAI-10 is a 10-item questionnaire to assess 1) subjective experience of drug and 2) attitudes and beliefs toward neuroleptics which may influence compliance in schizophrenia participants. It is the binary scale assessing the participant's subjective response. A 'compliant' response is scored as +1; a dysphoric response is scored as -1. A positive sum of items indicates a positive subjective response (SR); a negative sum of scores indicates a negative SR (non-compliant). The final score is the grand total of the positive and negative points. Total score ranges from (-) 10 to (+) 10, higher score indicates positive SR (compliant) and lower score indicates negative SR (non-compliant). Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 179 | 47 | 58
Units on a scale
  Baseline | 3.12 (4.65) | 3.49 (4.67) | 2.50 (4.88)
  Change at Week 24 | -0.46 (4.70) | -0.21 (4.92) | -1.00 (5.03)

10. Secondary Outcome: Change From Baseline in Symptom Checklist 90-R (SCL90-R) at Week 24
Description: The SCL90-R (Derogatis, 1992) measures 9 domains, including somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, which provides a global index of distress, the Global Severity Index (GSI). SCL-90-R includes 90 items rated on 5-point scale, ranging from 0 (not at all) to 4 (extremely). Total scale score range from 0 to 360. Higher scores indicate worsening of disease. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: The ITT population for efficacy included all the participants who received paliperidone ER at least once and who had at least 1 post baseline efficacy assessment. "N" (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 179 | 47 | 57
Units on a scale
  Baseline | 109.65 (67.00) | 107.23 (72.17) | 83.39 (60.41)
  Change at Week 24 | 2.42 (30.44) | 9.40 (32.31) | 1.16 (17.83)

11. Secondary Outcome: Change From Baseline in Krawiecka Scale Score at Week 24
Description: Psychopathology of participants was assessed by Krawiecka scale. Psychopathology of participants was assessed by Krawiecka scale, score ranges from 0 to 16. Higher score indicates worsening of disease. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 179 | 47 | 58
Units on a scale
  Baseline | 4.78 (3.12) | 3.45 (2.82) | 3.86 (2.96)
  Change at Week 24 | 0.94 (2.90) | 1.09 (2.80) | 1.09 (3.00)

12. Secondary Outcome: Change From Baseline in Total Personal and Social Performance (PSP) Score at Week 24
Description: The PSP scale assesses the degree of dysfunction within 4 domains of behavior: socially useful activities, personal and social relationships, self-care and disturbing and aggressive behavior. The score ranges from 1 to 100, divided into 10 equal intervals to rate the degree of difficulty (1, absent to 6, very severe) in each of the 4 domains. Participants with a score of 71 to 100 have a mild degree of difficulty; from 31 to 70, varying degrees of disability; less or equal to 30, functioning so poorly as to require intensive supervision. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 179 | 47 | 58
Units on a scale
  Baseline | 52.15 (15.44) | 57.91 (16.31) | 58.71 (12.62)
  Change at Week 24 | -6.50 (14.36) | -7.23 (12.49) | -6.28 (10.70)

13. Secondary Outcome: Change From Baseline in Sleep Quality Based on Visual Analog Scale at Week 24
Description: Sleep quality was assessed by an 11-point visual analog scale that rates how well participants slept. Participants indicated on the scale (from 0 to 100 millimeter) how well they slept in the previous 7 days (from 0: "very badly" to 100: "very well"). Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 179 | 47 | 58
Millimeter (mm)
  Baseline | 61.84 (29.34) | 71.55 (24.92) | 69.31 (23.48)
  Change at Week 24 | -0.84 (31.22) | -0.43 (30.25) | -0.67 (22.42)

14. Secondary Outcome: Change From Baseline in Daytime Drowsiness Based on Visual Analog Scale at Week 24
Description: Daytime drowsiness was assessed by an 11-point visual analog scale that rates how well participants slept. Participants indicated on the scale (from 0 to 100 millimeter) how often they felt drowsy in the previous 7 days (from 0: "very badly" to 100: "very well"). Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 179 | 47 | 58
Millimeter (mm)
  Baseline | 40.57 (31.79) | 45.96 (31.18) | 46.55 (28.65)
  Change at Week 24 | -1.18 (32.17) | 3.94 (28.02) | 10.05 (25.75)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 96
Description: Safety population included all the participants who received paliperidone extended-release (ER) at least once.
Arm/Group | Paliperidone
Serious Adverse Events (participants affected / at risk) | 21/289
Other Adverse Events (participants affected / at risk) | 112/289
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone (N=289)
Condition Aggravated (General disorders) | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1
Hepatic Enzyme Increased (Investigations) | 1
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Dystonia (Nervous system disorders) | 1
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Acute Psychosis (Psychiatric disorders) | 1
Completed Suicide (Psychiatric disorders) | 2
Delusion (Psychiatric disorders) | 1
Hallucination, Auditory (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 1
Psychotic Behaviour (Psychiatric disorders) | 2
Psychotic Disorder (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 4
Schizophrenia, Paranoid Type (Psychiatric disorders) | 1
Social Avoidant Behaviour (Psychiatric disorders) | 1
Suicidal Ideation (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone (N=289)
Constipation (Gastrointestinal disorders) | 11
Dry Mouth (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 8
Weight Increased (Investigations) | 6
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 7
Akathisia (Nervous system disorders) | 24
Bradykinesia (Nervous system disorders) | 12
Dizziness (Nervous system disorders) | 11
Dystonia (Nervous system disorders) | 9
Essential Tremor (Nervous system disorders) | 6
Extrapyramidal Disorder (Nervous system disorders) | 14
Headache (Nervous system disorders) | 10
Sedation (Nervous system disorders) | 6
Somnolence (Nervous system disorders) | 7
Tremor (Nervous system disorders) | 14
Insomnia (Psychiatric disorders) | 14

LIMITATIONS AND CAVEATS:
Some Adverse Events summaries were reported based on estimates due to the fact that they were not prepared in the original study report and the relevant definitions of the data elements were not available for these summaries to be regenerated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less